CLINICAL TRIAL: NCT06803095
Title: Efficacy of Walking Exercise With Dog on Tinnitus Complaints in Sleep Apnea
Brief Title: Efficacy of Walking Exercise With Dog on Tinnitus Complaints in Sleep Apnea (Obstructive Sleep Apnea)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ali Mohamed Ali ismail, Department of Physical Therapy for Cardiovascular/Respiratory Disorder and Geriatrics, Faculty of Physical Therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00014233-18
Record Dates: First submitted 2025-01-27; First posted 2025-01-31 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Tinnitus, Subjective; Obstructive Sleep Apnea
MeSH Terms: conditions — Tinnitus; Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group I (Experimental): the total participants of tinnitus (chronic subjective form) and obstructive sleep apnea (mild degree) in this group will be 20. This groups will follow low calorie diet.. this diet will be applied for 12 weeks.. during this period this group will receive free walking (30 min) with dog three timmes weekly.
  Interventions: Behavioral: free walking with dog and diet restriction
- Group II (Active Comparator): the total participants of tinnitus (chronic subjective form) and obstructive sleep apnea (mild degree) in this group will be 20. This group will follow low calorie diet only.. this diet will be applied for 12 weeks..
  Interventions: Behavioral: diet restriction

INTERVENTIONS:
Behavioral: free walking with dog and diet restriction — the total participants of tinnitus (chronic subjective form) and obstructive sleep apnea (mild degree) in this group will be 20. This group will follow low calorie diet.. this diet will be applied for 12 weeks.. during this period the study, this group will receive free walking (30 min) with dog three timmes weekly.
  Arms: group I
Behavioral: diet restriction — the total participants with tinnitus (chronic subjective form) and obstructive sleep apnea (mild degree) in this group will be 20. This group will follow low calorie diet only .. this diet will be applied for 12 weeks..
  Arms: Group II

SUMMARY:
there is evidence that tinnitus (chronic subjective form) is highly prevalent among patients with obstructive sleep apnea. exercise is recommneded in chronic subjective form) and obstructive sleep apnea. walking with dog increase adherence to walking to maintain continuity of physical activity

DETAILED DESCRIPTION:
the total participants will be forty in number.. those participants will complain form tinnitus (chronic subjective form) and obstructive sleep apnea (mild degree).. the particiapnts will divided to groups.. the number of subjects in each group will be 20. The groups (both groups) will follow low calorie diet.. this diet will be applied for 12 weeks.. during this period the study group will receive free walking (30 min) with dog three timmes weekly. the control group will not receive free walking with dog

ELIGIBILITY:
Inclusion Criteria:

* obese persons
* bilateral chronic subjective tinnitus
* mild obstructive sleep apnea (mild apnea hypopnea index)
* forty participants

Exclusion Criteria:

* body mass index more than 40 kg/m2.
* cardiovascular problems
* hepatorenal probelms
* autoimmune problems
* orthopedic probelms

Ages: 30 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — self-representation of gender identity.
Enrollment: 40 (Estimated)
Dates: Start 2024-12-12 (Actual); Primary Completion 2025-05-15 (Estimated); Study Completion 2025-05-15 (Estimated)

PRIMARY OUTCOMES:
tinnitus handicap inventory | it will be assessed after 12 weeks
  it is a questionaire assess tinnitus-associating life quality

SECONDARY OUTCOMES:
VAS of discomfort induced by tinnitus | it will be assessed after 12 weeks
  it is 10 com visual analogue scale
VAS of loudness of tinnitus | it will be assessed after 12 weeks
  it is 10 com visual analogue scale
apnea hyponea index | it will be assessed after 12 weeks
  it is number of occurrences of apnea and hyponea in hour
Eporwth sleepiness scale | it will be assessed after 12 weeks
  it will assess daytime sleepiness
Pittsburgh sleeping quality index | it will be assessed after 12 weeks
  it will assess sleep quality (subjective assessment)
Questionnaire of Depression, Anxiety, Stress Scales | it will be measured after 12 weeks
  it will contain 42 questions assessing psychological status (Depression, Anxiety, Stress) of participants
body mass index | it will be measured after 12 weeks
  it will be measured on empty stomach
wait circumference | it will be measured after 12 weeks
  it will be measured at umbilical level

CONTACTS AND LOCATIONS:
Overall Officials: Ali Ismail, lecturer, Principal Investigator — Cairo University
Locations (1):
- Cairo University, Dokki, Giza Governorate, Egypt